CLINICAL TRIAL: NCT05031078
Title: Assessing Immunological Basis of Durable Antibody Responses to 9-valent HPV Vaccination
Brief Title: Assessing Durable Antibody Response to HPV Vaccination
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Erin Scherer, PhD, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002830
Record Dates: First submitted 2021-08-27; First posted 2021-09-01 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: HPV
Keywords: HPV
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Lymph node sampling at D-30 to D0, D14 and D30 (Experimental): Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180.
  Group 1 will undergo an FNA at D-30 to D0. Participants will repeat the procedure at D14±5 and D30±5.
  Bone marrow sampling will be done for all groups at D730 and D1825.
  Interventions: Biological: Gardasil-9; Drug: Lidocaine injections
- Group 2: Lymph node sampling at D60, D74 and D90 (Experimental): Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180.
  Participants will undergo an FNA on the same day, but prior to, the second vaccine dose (D60±5; Visit 8) or up to 5 days before. Participants will repeat the procedure at Visit 8 + 14±5 days and Visit 8 + 30±5 days.
  Bone marrow sampling will be done for all groups at D730 and D1825.
  Interventions: Biological: Gardasil-9; Drug: Lidocaine injections
- Group 3: Lymph node sampling at D180, D194 and D210 (Experimental): Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180.
  Group 3 will undergo an FNA on the same day, but prior to, the third vaccine dose (D180±5; Visit 13) or up to 5 days before. Participants will repeat the procedure at Visit 13 + 14±5 days and Visit 13 + 30±5 days.
  Bone marrow sampling will be done for all groups at D730 and D1825.
  Interventions: Biological: Gardasil-9; Drug: Lidocaine injections

INTERVENTIONS:
Biological: Gardasil-9 — Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180 The 9-valent HPV vaccine, or Gardasil-9, is a non-infectious recombinant vaccine prepared from the purified virus-like particles (VLPs) of the major capsid (L1) protein of HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58.
  Gardasil-9 is supplied as a 0.5-mL single-dose vial or 0.5-mL single-dose prefilled Luer Lock syringe with tip cap.
  Other Names: HPV vaccine
Drug: Lidocaine injections — 1-2% lidocaine injections.
  1% lidocaine, an FDA approved local anesthetic, will be injected subcutaneously to numb the area of the lymph node being sampled; whereas 1-2% lidocaine will be injected into the tissue surrounding the area where the bone marrow will be removed. In adults the recommended dose is 7 mg/kg with a maximum of 500 mg.

SUMMARY:
This is a single center, longitudinal cohort study in which subjects will receive 9-valent HPV vaccine according to package insert (i.e., one dose of 9-valent HPV vaccine on day (D) 0 followed by a second dose 2 months later and a third dose 6 months later).

Immune responses in the blood, saliva, bone marrow, and lymph nodes will be assessed in subjects receiving the HPV vaccine.

Blood samples for immunologic testing will be collected at screening (from D-60 to D-45), on D0 (before vaccination), D1 (optional visit), D7±1, D14±5, D30±5, D60±5 (Visit 8, before vaccination), Visit 8 +1 day (optional visit), Visit 8 + 7±1 days, Visit 8 + 14±5 days, Visit 8 + 30±5 days, D180±5 (Visit 13, before vaccination), Visit 13 + 7±1 days, Visit 13 + 14±5 days, Visit 13 + 30±5 days, D365±14, D730±14, D1095±14, D1460±14, D1825±30. Saliva samples for antibody testing will be collected on D0 (before vaccination), D30, D60 (before vaccination), Visit 8 + 30±5 days, D180 (before vaccination), Visit 13 + 30±5 days, D365, and D730.

Axillary lymph node sampling by fine needle aspiration will be done 3 times per group. Group 1 will have lymph node sampling done D-30 to D0, D14, and D30. Group 2 will have lymph node sampling done D60, Visit 8 + 14±5 days, and Visit 8 + 30±5 days. Group 3 will have lymph node sampling D180, Visit 13 + 14±5 days, and Visit 13 + 30±5 days. Bone marrow sampling will be done for all groups at D730±14 and D1825±30.

DETAILED DESCRIPTION:
Human papillomaviruses (HPV) cause cervical, anal, oropharyngeal, vulvar, vaginal, and penile cancers. There are over 200 types of HPV; 12 are known to cause cancer. The current HPV vaccine is a subunit vaccine, meaning it is made of only part of the virus (a protein) and cannot infect humans. The HPV vaccine is highly effective at preventing disease by HPV types that cause 90% of cancer cases and 90% of genital warts cases in women and men who do not have ongoing or prior HPV infection.

Most vaccines protect by generating antibodies. Importantly, the HPV vaccine, first approved in 2006, has been shown to make high levels of antibodies against HPV that last for >10 years. The durability of HPV vaccine antibody levels is exceptional compared to other approved and experimental subunit vaccines whose antibody levels drop more rapidly. However, how the HPV vaccine - let alone any vaccine - generates long-lasting antibodies is not understood. Understanding how vaccines make high levels of long-lasting antibodies will help the efforts to successfully and reliably design new vaccines that make these highly desired responses (like vaccines against new pandemics).

The investigators designed this study to better understand how the HPV vaccine generates such high levels of long-lasting antibodies in humans. To do this, the investigators need to study early immune responses in lymph nodes, which is where cells that make antibodies (B cells) are activated by the vaccine. The investigators will also need to study immune responses in blood. For example, to measure the levels of antibodies in blood and also the levels of cells that help B cells (helper T cells). As the HPV vaccine can protect against oropharyngeal cancer, the study team aim to understand the level of antibodies in the saliva and how the antibodies compare to blood. Finally, antibodies themselves are not long-lived as proteins, but the cells that make these antibodies are (specialized B cells called plasma cells). Plasma cells are found in the bone marrow. It is important that the research team finds and study these cells making antibodies against HPV, so the investigators can better understand how they contribute to long-lasting antibody levels.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-45 years old (inclusive), as the HPV vaccine is approved for this age range in adults
* BMI ≤ 32.
* Able to understand and give informed consent (provided in American English).
* Must be in good health based on physical examination, vital signs, medical history, and the investigator's clinical judgment.
* Must be available and willing to participate for the duration of this study
* Must be willing to undergo lymph node fine needle aspiration and bone marrow aspiration
* Must be willing to consent to the future use of remaining (residual) samples/specimens.

Exclusion Criteria:

* Ever received a dose of an HPV vaccine
* HPV 6, 11, 16, 18, 31, 33, 45, 52 or 58 seropositivity
* Any history of genital warts, an abnormal pap smear, or positive HPV DNA test
* Has known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products
* Has known allergy or history of anaphylaxis to yeast or products containing yeast
* Any allergy to lidocaine.
* Pregnancy or breast feeding.
* Subjects who believe they cannot tolerate the lymph node fine needle aspirate or bone marrow aspirate procedures without sedation
* Any history of lymphoma involving axillary nodes, any history of breast cancer, bilateral inflammatory process of upper arms in the past 2 weeks, prior breast or axillary biopsy and/or surgery that in the opinion of the investigator would affect the immune response results.
* Local infection, lymphadenitis, or rash in targeted area.
* Received any vaccine from 14 days before vaccine dose until 30 days after each vaccine dose.*

  *An individual who is initially excluded from study participation based on one or more of the time-limited exclusion criteria (fever, receipt of other vaccines) may be reconsidered for enrollment once the condition has resolved as long as the subject continues to meet all other entry criteria.
* Volunteers with fever (≥100.4 F or 38°C regardless of the route) within 3 days prior to vaccination.*

  *An individual who is initially excluded from study participation based on one or more of the time-limited exclusion criteria (fever, receipt of other vaccines) may be reconsidered for enrollment once the condition has resolved as long as the subject continues to meet all other entry criteria.
* History of or presence of severe co-morbidities as determined by the investigator, including autoimmune disease, or clinically significant cardiac, pulmonary, gastrointestinal, hepatic, rheumatologic, renal disease, thrombocytopenia, and grade 4 hypertension*.

  *Grade 4 hypertension per CTCAE criteria is defined as Life-threatening consequences (e.g., malignant hypertension, transient or permanent neurologic deficit, hypertensive)
* History of a bleeding disorder or currently taking anti-coagulant products* (e.g. warfarin, direct thrombin inhibitors, heparin products, etc.), anti-platelet products, and/or NSAIDs including aspirin.

  *including in the past week; however, an individual who is initially excluded from study participation based on one or more of the time-limited exclusion criteria may be reconsidered for enrollment once the condition has resolved as long as the subject continues to meet all other entry criteria
* Has history of active malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure.
* Current and/or expected immunosuppression due to cancer, receipt of chemotherapy, radiation therapy, and any other immunosuppressive therapies (including anti-TNF therapy).
* Has known or suspected congenital or acquired immunodeficiency, including functional or anatomic asplenia, or recent history or current use of immunosuppressive therapy*.

  *Anti-cancer chemotherapy or radiation therapy within the preceding 3 years, or long-term (≥2 weeks within the previous 3 months) systemic corticosteroid therapy (e.g., prednisone at a dosage of ≥20 mg per day or on alternative days). Intranasal or topical prednisone (or equivalent) are allowed.
* Known chronic infections including, but not limited to, known HIV, tuberculosis, hepatitis B or C.
* Is post-organ, bone marrow, and/or stem cell transplant, whether or not on chronic immunosuppressive therapy.
* Received blood products or immunoglobulin in the 3 months before study entry or planned use during this study.
* Had major surgery (per the investigator's judgment) within 4 weeks before study entry or planned major surgery during this study.
* Insulin-dependent diabetes* mellitus type 1 or type 2 requiring therapy

  *History of isolated gestational diabetes is not an exclusion criterion.
* Received experimental therapeutic agents within 12 months before first vaccine dose or plans to receive any experimental therapeutic agents 12 months after first vaccine dose that, in the opinion of the investigator, would interfere with the safety or objectives of the study. COVID-19 vaccines that fall under FDA EUA will be treated as approved vaccines for the purposes of this study.
* Is currently participating or plans to participate in another clinical study which would involve receipt of an investigational product or undergo a procedure that, in the opinion of the investigator, would interfere with safety or objectives of the study.
* Current diagnosed or self-reported alcohol abuse, drug abuse, or psychiatric conditions that in the opinion of the investigator would preclude compliance with the study.
* Social, occupational, or any other condition that in the opinion of the investigator might interfere with compliance with the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2026-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Scherer, Ph.D., Principal Investigator — Emory University
Locations (2):
- United States (2):
  - The Hope Clinic of Emory University, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, after deidentification, and RNA sequencing data
Time Frame: Available immediately following publication. No end date.
Access Criteria: De-identified data will be published in an open access journal with no access restrictions; De-identified RNA Seq data will be deposited at NCBI/ Gene Expression Omnibus or similar public database with no access restrictions

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Lymph Node Sampling at D-30 to D0, D14 and D30: Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180.
  Group 1 will undergo an FNA at D-30 to D0. Participants will repeat the procedure at D14±5 and D30±5.
  Bone marrow sampling will be done for all groups at D730 and D1825.
  Gardasil-9: Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180.
  The 9-valent HPV vaccine, or Gardasil-9, is a non-infectious recombinant vaccine prepared from the purified virus-like particles (VLPs) of the major capsid (L1) protein of HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58.
  Gardasil-9 is supplied as a 0.5-mL single-dose vial or 0.5-mL single-dose prefilled Luer Lock syringe with tip cap.
  Lidocaine injections: 1-2% lidocaine injections.
  1% lidocaine, an FDA approved local anesthetic, will be injected subcutaneously to numb the area of the lymph node being sampled; whereas 1-2% lidocaine will be injected into the tissue surrounding the area where the bone marrow will be removed. In adults the recommended dose is 7 mg/kg with a maximum of 500 mg.
- Group 2: Lymph Node Sampling at D60, D74 and D90: Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180.
  Participants will undergo an FNA on the same day, but prior to, the second vaccine dose (D60±5; Visit 8) or up to 5 days before. Participants will repeat the procedure at Visit 8 + 14±5 days and Visit 8 + 30±5 days.
  Bone marrow sampling will be done for all groups at D730 and D1825.
  Gardasil-9: Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180.
  The 9-valent HPV vaccine, or Gardasil-9, is a non-infectious recombinant vaccine prepared from the purified virus-like particles (VLPs) of the major capsid (L1) protein of HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58.
  Gardasil-9 is supplied as a 0.5-mL single-dose vial or 0.5-mL single-dose prefilled Luer Lock syringe with tip cap.
  Lidocaine injections: 1-2% lidocaine injections.
  1% lidocaine, an FDA approved local anesthetic, will be injected subcutaneously to numb the area of the lymph node being sampled; whereas 1-2% lidocaine will be injected into the tissue surrounding the area where the bone marrow will be removed. In adults the recommended dose is 7 mg/kg with a maximum of 500 mg.
- Group 3: Lymph Node Sampling at D180, D194 and D210: Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180.
  Group 3 will undergo an FNA on the same day, but prior to, the third vaccine dose (D180±5; Visit 13) or up to 5 days before. Participants will repeat the procedure at Visit 13 + 14±5 days and Visit 13 + 30±5 days.
  Bone marrow sampling will be done for all groups at D730 and D1825.
  Gardasil-9: Participants will receive 3 doses of 9-valent HPV vaccine (Gardasil 9) at D0, D60, and D180.
  The 9-valent HPV vaccine, or Gardasil-9, is a non-infectious recombinant vaccine prepared from the purified virus-like particles (VLPs) of the major capsid (L1) protein of HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58.
  Gardasil-9 is supplied as a 0.5-mL single-dose vial or 0.5-mL single-dose prefilled Luer Lock syringe with tip cap.
  Lidocaine injections: 1-2% lidocaine injections.
  1% lidocaine, an FDA approved local anesthetic, will be injected subcutaneously to numb the area of the lymph node being sampled; whereas 1-2% lidocaine will be injected into the tissue surrounding the area where the bone marrow will be removed. In adults the recommended dose is 7 mg/kg with a maximum of 500 mg.
Period: Overall Study
Arm/Group | Group 1: Lymph Node Sampling at D-30 to D0, D14 and D30 | Group 2: Lymph Node Sampling at D60, D74 and D90 | Group 3: Lymph Node Sampling at D180, D194 and D210
Started | 8 | 5 | 4
Completed | 8 | 4 | 4
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Lymph Node Sampling at D-30 to D0, D14 and D30 | Group 2: Lymph Node Sampling at D60, D74 and D90 | Group 3: Lymph Node Sampling at D180, D194 and D210 | Total
Number analyzed (Participants) | 8 | 5 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (5.3) | 29.4 (6.4) | 32.2 (7.8) | 34.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 7
  Male | 4 | 4 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 7 | 5 | 2 | 14
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Minimum Four-fold Rise in Post-vaccination HPV-16 and HPV-18 Neutralizing Antibody Titers
Description: Determining the number of participants with a minimum four-fold rise in post-vaccination HPV-16 and HPV-18 neutralizing antibody titers determined using an HPV pseudovirus neutralization assay
Time Frame: 30 days after receiving the third and final vaccine dose (approximately Day 210 after first vaccine dose)
Population: Participants that completed the primary outcome (n = 16) were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Lymph Node Sampling at D-30 to D0, D14 and D30 | Group 2: Lymph Node Sampling at D60, D74 and D90 | Group 3: Lymph Node Sampling at D180, D194 and D210
Number analyzed (Participants) | 8 | 4 | 4
Participants | 8 | 4 | 4

2. Secondary Outcome: Change in Number of HPV-specific Memory B Cell (Bmem) Response From Baseline
Description: Magnitude of HPV specific Bmem responses will be assessed at baseline and following 9-valent HPV vaccination
  Baseline (Day 0), Day 30, Day 180, Day 210, Day 365, Day 730
Time Frame: Baseline (Day 0), Day 30, Day 180, Day 210, Day 365, Day 730 post-intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data collected between time of consent and 30 days after receiving the third and final vaccine dose (approximately Day 210).
Arm/Group | Group 1: Lymph Node Sampling at D-30 to D0, D14 and D30 | Group 2: Lymph Node Sampling at D60, D74 and D90 | Group 3: Lymph Node Sampling at D180, D194 and D210
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2025-05-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT05031078/Prot_001.pdf